CLINICAL TRIAL: NCT01762553
Title: TEA (Together for Empowerment Activities)for Families and Children: A Randomized Intervention Trial
Brief Title: TEA for Families and Children: A Randomized Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Li Li, Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HD068165-01 (NIH)
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Behaviors; Health
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): The TEA intervention program will be implemented for the intervention group. The TEA intervention has three modules (healthy body & healthy mind, family interaction, and quality of life) logically connected to each other and implemented at three levels from individual, family to the community: 1) TEA Gathering is a small group training session for PLH and their family members to deal with HIV-related challenges at individual level; 2) TEA Time is home based family activities for PLHs and their family members to interact with their children after each TEA Gathering to promote family positive interaction; 3) TEA Garden is the community events that built social integration for HIV affected families to live a healthy social life and to build sustained, supportive relationships in their communities. There will be reunions once a month for 12 months after the completion of the TEA intervention.
  Interventions: Behavioral: The TEA intervention
- Control (No Intervention): In order to tease out the impact of the proposed intervention from the impact of attention in general, we will add limited activities to the control group condition. The differences between the intervention and control conditions consist in both contents and formats. For the control group, there will only be group sessions once a week for three weeks starting after baseline assessment. The content of the sessions for the control group will focus on basic care, health education and promotion, nutrition, personal and family hygiene. The Essential Care Package (ECP), a set of education materials originally developed by the World Health Organization (WHO) and supported by the Global Fund Project, will be used and explained in these group sessions. Health workers from villages in the control group will also visit participating families once a week for the initial three weeks and once a month for 12 months.

INTERVENTIONS:
Behavioral: The TEA intervention — TEA Gathering is a small group training session for PLH and their family members to deal with HIV-related challenges at individual level; TEA Time is home based family activities for PLHs and their family members to interact with their children after each TEA Gathering to promote family positive interaction; TEA Garden is the community events that built social integration for HIV affected families to live a healthy social life and to build sustained, supportive relationships in their communities. There will be reunions once a month for 12 months after the completion of the TEA intervention.
  Arms: intervention

SUMMARY:
The impact of HIV/AIDS is negatively influencing the affected families and their next generation. HIV is radiating through the extended families, shifting the life patterns not only for the parents living with HIV/AIDS (PLH), but also for their children, partners, and other family members. To help PLHs and their family members, the TEA intervention has been developed, refined and piloted in the previous study. The goal of this study is to implement the TEA intervention in a full scale to determine its efficacy and the potential for enhancing HIV policy and programs that support HIV-affected families to cope with the challenges in China in responding to the global HIV epidemic.

DETAILED DESCRIPTION:
This 5-year project is a randomized controlled trial of the TEA (Together for Empowerment Activities) intervention, a family intervention for HIV-affected families in rural areas of China.

The impact of HIV/AIDS is negatively influencing the affected families and their next generation. Currently in China, there are about 740,000 families living with HIV and 105,000 of them have developed AIDS. HIV is radiating through the extended families, shifting the life patterns not only for the parents living with HIV/AIDS (PLH), but also for their children, partners, and other family members. The negative impact of HIV is compounded by Chinese tradition of accepting illness stoically and not discussing difficult issues within the family due to shame and fear. Chronic illness also reverses the Chinese traditional family roles especially when the ill parents are not capable of contributing to housework or providing financial stability and the further burden rests on the children. As a result, the relationship between parents, family members and children is significantly strained. To help PLHs and their family members, the TEA intervention has been developed, refined and piloted in the previous study. The goal of this study is to implement the TEA intervention in a full scale to determine its efficacy and the potential for enhancing HIV policy and programs that support HIV-affected families to cope with the challenges in China in responding to the global HIV epidemic.

TEA intervention will have six sessions (plus a preparation session) delivered at three levels simultaneously: 1) TEA Gathering (small group for PLH and their family members), 2) TEA Time (home-based family activities with children that accompany each TEA Gathering), and 3) TEA Garden (community events that build social integration). Built on the successful pilot work by the collaborative team, this intervention trial will include 24 administrative villages with 20 families each, resulting in a total of 480 participating families affected by HIV. The administrative villages will be randomized into two groups (12 villages in each): TEA intervention group and control group (with 240 families in each group). A total of 240 PLH, 240 family members and 360 children at age of 6-18 will be recruited in each group. After the baseline assessment, the TEA intervention will be conducted in the intervention group, but not in the control group. Follow-up assessments will be conducted at 6, 12, 18 and 24 months after the intervention is delivered. The impact of the intervention will be assessed by comparing the outcomes measures at baseline and 6-, 12-, 18- and 24-month follow-ups between the intervention and control groups for HIV-affected families, including PLH, family members, and children in poor, rural areas in China (Figure 1). The primary outcomes are children's health, mental health, and behavioral adjustment. The secondary outcomes will be the PLH's and family members' physical health, mental health, and quality of life, as well as family indicators such as family daily routines, positive interactions, parenting, coping, and community integration.

The study will be implemented in Anhui, China. Four counties, Lixin, Funan, Yinzhou and Linquan in Anhui Province have been selected as project sites based on the sample size of HIV-affected families and similarity of demographics. Within the selected counties, the administrative villages that have 20 or more HIV-affected families with at least one child aged 6-18 have been identified based on the current epidemiological data, resulting in a total of 24 villages for this study. Through a randomization procedure, 12 villages will be randomized to TEA intervention group and 12 villages to control group. Only the families that have one PLH, at least one family member, and at least one child aged at 6-18 years will be invited to participate. We will recruit all families from each of the villages, resulting in a total of about 480 HIV-affected families with 480 PLHs, 480 family members and 720 children.

The purpose of this study is to develop a feasible and practical intervention strategy through a randomized controlled intervention trial, which will help HIV-affected families in rural areas of China to face the challenges of HIV and improve their health and quality of life.

The Specific Aims of the study are:

1. To test that the children in the intervention group, compared to those in the control group, will have significantly better physical health, mental health, and behavioral outcomes.
2. To test that the PLH and family members in the intervention group, compared to those in the control group, will have significantly improved physical health, mental health, and quality of life outcomes.
3. To investigate how outcomes of the children, PLH, and family members are mediated by family indicators such as consistent daily routines, positive family interactions, parenting, coping, and community integration.

ELIGIBILITY:
Inclusion Criteria:

* PLH: age 18 or over, being a resident of one of the 24 selected villages, who is currently HIV sero-positive parent of a child between 6-18 years in his/her family, and who provide informed consent.
* Family members: 18 years and older, being a resident of one of the 24 selected villages, who is aware of PLH's HIV status, who has consent from participating PLH to be invited to join the study, and who provides informed consent. If there are two PLHs in a household, they both will be recruited as PLH participants.
* Children: aged 6-18 years, being a resident of one of the 24 selected villages, who lives in a HIV-affected family in which at least one or both parents is HIV-positive, and who provides parent/guardian permission, child/youth assent forms or informed consent if aged 18.

Exclusion Criteria:

Those who cannot give informed consent (e.g., intoxicated) Those who have a permanent disability (e.g., deaf, serious mental illness, mental retardation).

Anyone who does not meet the inclusion criteria.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1533 (Actual)
Dates: Start 2011-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
children's behavior problems and health | Change from baseline to 6-, 12-, 18-, and 24 month follow up
  During the intervention pilot, we conducted assessments for children aged 6-12 and 13-18, respectively. We also asked adults questions regarding their children's behavior. Health for children will be assessed by the questions from the China Global School-Based Student Health Survey.50 Questions from the China Children Health and Nutrition Survey will be filled out by PLH. Mental health will be measured by the Everyday Stress Index (α=0.79), and the Rosenberg Self-Esteem Scale54 (α=0.69). For children aged 13-18, the Emotional Quotient Scale (α=0.69) including subscales of motivation, relationship, and satisfaction will be administered. Behavioral adjustment will be measured by their self reports on school performance and satisfaction, consistent family routines (α=0.60), peer relations, and delinquent behaviors (α=0.70).

SECONDARY OUTCOMES:
People living with HIV and Family member | Change from baseline to 6-. 12-, 18-, and 24 month follow up
  Health of the PLH and FM will be assessed by using the Medical Outcomes Study (MOS)-HIV for PLH and MOS-Short Form-36 (SF-36) for family members. For PLH's health, MOS-HIV physical functioning (α=0.85), pain, energy/fatigue (α=0.85), and health distress (α=0.72) will be used. For FMs' health, MOS-SF36 will be used (α=0.89). Mental health of PLH will be assessed using MOS-HIV mental health scale (α=0.84) and cognitive functioning scale (α=0.65). For both PLH and FM, Zung Self-Rating Depression Scale will be used to assess their level of depressive symptoms. This instrument has been used by our team twice in the pilot studies (α=0.80 for PLH and α=0.83 for FM). PTSD will be measured by a brief 7-item scale (α=0.77) for PLH only. FM burden will be assessed with the Perceived Caregiver Burden Scale (PCB). Quality of life of PLH will be assessed using MOS-HIV general health perceptions (α=0.81) and role functioning (α=0.79).

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, PhD, Principal Investigator — NPI-Center for Community Health, UCLA
Locations (1):
- Anhui Provincial Center for Disease Control and Prevention, Hefei, Anhui, China

REFERENCES:
- [Derived] Li L, Liang LJ, Lin C, Lan CW, Ji G, Xiao Y. Changes in behavioral outcomes among children affected by HIV: Results of a randomized controlled trial in China. J Health Psychol. 2019 Sep;24(11):1581-1594. doi: 10.1177/1359105317746479. Epub 2017 Dec 15. PMID 29243519
- [Derived] Li L, Ji G, Liang LJ, Lin C, Hsieh J, Lan CW, Xiao Y. Efficacy of a multilevel intervention on the mental health of people living with HIV and their family members in rural China. Health Psychol. 2017 Sep;36(9):863-871. doi: 10.1037/hea0000503. Epub 2017 May 22. PMID 28530433